CLINICAL TRIAL: NCT00855634
Title: Extended Versus Standard Resection in Two Cohorts of Patients With Adenocarcinoma of the Pancreas: Minimal Metastatic Disease or Venous Infiltration - a Randomized Trial
Brief Title: Resection in Pancreatic Cancer With Minimal Metastatic Disease or Venous Infiltration Trial at Technische Universität München
Acronym: PaMeViTUM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol planned interim analysis after two years showed very low recruitment in cohort 1 and low recruitment in cohort 2.
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUM-Chir-001/2009
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2009-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; metastasis; venous infiltration; Pancreatic cancer with minimal metastatic disease or venous infiltration
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): COHORT 1 (minimal metastatic disease):
  * Arm 1 (intervention): resection of the primary tumor, followed by resection of the liver metastasis/metastases
  * Arm 2 (control): exploration and/or gastroenterostomy and/or hepaticojejunostomy/choledochojejunostomy
  Interventions: Procedure: Resection of metastases
- 2 (Active Comparator): COHORT 2 (venous infiltration):
  * Arm 1 (intervention): resection of the primary tumor with resection of the portal vein (and/or superior mesenteric vein/splenic vein (SMV/SV)
  * Arm 2 (control): resection of the primary tumor with dissection of the portal vein (and/or superior mesenteric vein/splenic vein (SMV/SV) plus tumor masses adjacent to these veins; no venous resection
  Interventions: Procedure: Resection of infiltrated veins

INTERVENTIONS:
Procedure: Resection of metastases — resection of the primary tumor, followed by resection of the liver metastasis/metastases
  Arms: 1
Procedure: Resection of infiltrated veins — resection of the primary tumor with resection of the portal vein (and/or superior mesenteric vein/splenic
  Arms: 2

SUMMARY:
PaMeViTUM is a mono-centric prospective randomized controlled trial that compares different operating procedures in patients with pancreatic cancer and minimal metastatic disease or venous infiltration.

DETAILED DESCRIPTION:
PaMeViTUM is a mono-centric prospective randomized controlled trial comparing different operating procedures in patients with pancreatic cancer and minimal metastatic disease or venous infiltration. Patients will be randomized intraoperatively after fulfilling all inclusion criteria (in particular: suspicion of cancer of the pancreas and an intraoperative histologically proven diagnosis of pancreatic adenocarcinoma; intraoperative assessment of tumor as potentially locally respectable). If no metastases and no infiltration of the portal vein are detected during the operation, the standard resection will be performed (for tumors of the pancreatic head: (pylorus-preserving) pancreaticoduodenectomy; for tumors of the pancreatic body/tail: distal (left) pancreatic resections; for tumors of the head and body/tail: total pancreatectomy). In the case of tumor infiltration of the pyloric region or the distal stomach, a classical pancreaticoduodenectomy will be performed.

If the patient has pancreatic cancer with minimal metastatic disease (COHORT 1) and fulfills all inclusion criteria, she/he will be randomized into one of the following arms:

* Arm 1 (intervention): resection of the primary tumor, followed by resection of the liver metastasis/metastases
* Arm 2 (control): exploration and/or gastroenterostomy and/or hepaticojejunostomy/choledochojejunostomy

If there are no liver metastases, following mobilization (and potentially also the dissection of the pancreas at the pancreatic head), the extension of the tumor towards the superior mesenteric/splenic/portal vein is examined. If there is venous infiltration (COHORT 2) and the patient fulfills the inclusion criteria, she/he will be randomized into one of the following arms:

* Arm 1 (intervention): resection of the primary tumor with resection of the portal vein (and/or superior mesenteric vein/splenic vein (SMV/SV)
* Arm 2 (control): resection of the primary tumor with dissection of the portal vein (and/or superior mesenteric vein/splenic vein (SMV/SV) plus tumor masses adjacent to these veins; no venous resection The aim of this study is to demonstrate that an extension of the resectability criteria in patients with pancreatic cancer and 1) minimal metastatic disease OR 2) venous infiltration improves overall survival. A secondary aim of the study is to prove that resection in these patient cohorts improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of cancer of the pancreas and an intraoperative histologically proven diagnosis of pancreatic adenocarcinoma.
* intraoperative assessment of tumor as potentially locally resectable
* COHORT 1: Minimal metastatic disease
* COHORT 2: Venous infiltration
* ability to sign the informed consent.
* Karnofsky performance status > 70.
* Life-expectancy of more than 3 months.
* able to attend follow-up.
* no previous or concurrent malignancy diagnoses, except non-melanoma skin cancer and in situ carcinoma of the cervix.
* no serious medical, psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up.
* patients older than 18 years.
* no pregnant or lactating women.
* preoperative evaluation by thin-sliced CT scans with:
* No evidence of substantial extra-pancreatic disease, i.e. no evidence of malignant ascites, extended liver metastasis (>5 metastatic lesions), spread to other distant abdominal organs, peritoneal metastasis, spread to extra-abdominal organs.
* No evidence of extension of the tumor into the celiac axis or superior mesenteric artery (T4 disease).
* intraoperative findings with:
* tumor assessed as potentially locally resectable.
* no signs of peritoneal metastasis or tumor manifestations outside of the pancreas and the liver.
* frozen section: adenocarcinoma

Exclusion Criteria:

* extrapancreatic disease (except minimal metastatic disease of the liver, see above)
* concomitant venous infiltration and minimal metastatic disease
* extension of the tumor into the celiac axis or superior mesenteric artery
* life expectancy of less than 3 months
* previous or concurrent malignancy diagnosis, except non-melanoma skin cancer and in situ carcinoma of the cervix
* conditions potentially hampering compliance (also inclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2009-08; Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Quality of life Perioperative morbidity and mortality 1-year survival and 2-year survival | Additional 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery and Institute of Statistics Klinikum rechts der Isar der Technischen Universität München Ismaningerstrasse 22 81675 München, Germany, München, Germany

REFERENCES:
- [Derived] Argentiero A, Calabrese A, Sciacovelli AM, Delcuratolo S, Solimando AG, Brunetti O. Complete Response of Synchronous Liver Metastasis in a Pancreatic Ductal Adenocarcinoma, When Surgery Could Represent a Therapeutic Option. Can J Gastroenterol Hepatol. 2020 Oct 9;2020:8679751. doi: 10.1155/2020/8679751. eCollection 2020. PMID 33102398